CLINICAL TRIAL: NCT06735703
Title: Incidince of PROM with GBS Infection and Prophylaxis Against It
Brief Title: Group B Streptococcus Infection and PROM Incidince
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Kamel, Dina mohamedkamel, Assiut University
Other Study IDs: GBS WITH PROM
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Premature Rupture of Fetal Membranes; Group B Streptococcal Infection
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Streptococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women after 34 wks with PROM
  Interventions: Drug: To provide ampicillin sulbactam to pregnant women with premature rupture of membrane

INTERVENTIONS:
Drug: To provide ampicillin sulbactam to pregnant women with premature rupture of membrane — To provide ampicillin sulbactam tonpregnant women with premature rupture of membrane after 34 wks gestation

SUMMARY:
To investigate incidince of prom with GBS infection and role of prophylaxis against it

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with prom after 34 wks festation

Exclusion Criteria:

* Bleeding disorder
* emergency conditions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with prom
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-12-09 (Estimated); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Incidince of prom with GBS infection and prophylaxis against it | Baseline